CLINICAL TRIAL: NCT01638234
Title: Effectiveness of Melatonin Supplement in the Management of Sleep Disturbances in Children With Atopic Dermatitis
Brief Title: Effectiveness of Melatonin for Sleep Disturbances in Children With Atopic Dermatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200902026M
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Starch pill (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Melatonin (Experimental)
  Interventions: Dietary Supplement: Melatonin

INTERVENTIONS:
Dietary Supplement: Melatonin — melatonin 3 mg tab 1 tab po hs for 4 weeks
  Arms: Melatonin
Dietary Supplement: Placebo — starch pill
  Arms: Starch pill

SUMMARY:
Sleep disturbance is a common complaint among patients with atopic dermatitis(AD). Melatonin may aid sleep and also has anti-inflammatory properties, and has been suggested in managing sleep disturbance in AD patients. However, there has been no large randomized controlled trials. Hence the objective of this double-blind randomized controlled study is to determine whether supplementing melatonin is effective in improving sleep problems in children with AD.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 and 18 years of age with mild to moderate AD, affecting at least 5% of total body surface area, and with sleep problems in the previous 3 months

Exclusion Criteria:

1. Those who had failed other systemic and/or topical immunosuppressive agents such as tacrolimus, methotrexate, or cyclosporine
2. Those who had received therapy for insomnia within 4 weeks before the baseline visit
3. Those who were, in the opinion of the investigator, known to be unreliable or noncompliant with medical treatment or appointments
4. Those who had drug abuse problems, mental health dysfunction, or other factors limiting their ability to cooperate fully
5. Those who were taking antihistamines, oral immunosuppressant medication, or antidepressant medication
6. Pregnant and lactating women and those who are presently planning to get pregnant
7. Those who had any other condition or earlier/current treatment which, in the opinion of the investigator, would render the participant ineligible for the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Objective sleep measures as measured by actigraphs and SCORAD | 4 weeks
  actigraph parameters including sleep latency, sleep efficiency, total sleep time, and wake episodes and duration; SCORAD and objective SCORAD for disease severity assessment

SECONDARY OUTCOMES:
urine and serum cytokines | 4 weeks
  serum levels of melatonin, urinary levels of 6-hydroxymelatonin sulfate, and serum levels of cytokines associated with sleep regulation including IL-10, IL-6, IL-4, IL-1b, and IL-31
total and allergen-specific IgE | 4 weeks
  total serum IgE and allergen specific IgE to Derp, Derf, SEA, and SEB
sleep parameters measured by polysomnography | 4 weeks
  sleep onset latency, sleep efficiency, wake episodes and duration, total sleep time, sleep stages, limb movement index
subjective improvement in symptoms | 4 weeks
  subjective assessment of whether sleep and dermatitis improved after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Hong Lee, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chang YS, Lin MH, Lee JH, Lee PL, Dai YS, Chu KH, Sun C, Lin YT, Wang LC, Yu HH, Yang YH, Chen CA, Wan KS, Chiang BL. Melatonin Supplementation for Children With Atopic Dermatitis and Sleep Disturbance: A Randomized Clinical Trial. JAMA Pediatr. 2016 Jan;170(1):35-42. doi: 10.1001/jamapediatrics.2015.3092. PMID 26569624